CLINICAL TRIAL: NCT02608840
Title: Auditory Stimulation of Slow Wave Sleep and Memory in Mild Cognitive Impairment and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roneil Malkani, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00200555
Record Dates: First submitted 2015-11-06; First posted 2015-11-20 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment
Keywords: slow-wave sleep; cognition; auditory stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MCI auditory stimulation (Experimental): MCI patients receiving auditory stimulation during sleep (crossover arm 1)
  Interventions: Other: Auditory stimulation during sleep
- MCI sham stimulation (Sham Comparator): Sham intervention: MCI patients sleeping with headphones but sounds not played (crossover arm 2)
  Interventions: Other: Sham Intervention
- Older adult auditory stimulation (Experimental): healthy older adults receiving auditory stimulation during sleep (crossover arm 1)
  Interventions: Other: Auditory stimulation during sleep
- older adult sham stimulation (Sham Comparator): Sham intervention: healthy older adults sleeping with headphones but sounds not played (crossover arm 2)
  Interventions: Other: Sham Intervention

INTERVENTIONS:
Other: Auditory stimulation during sleep — The intervention is a brain computer interface program which measures brain electroencephalogram to identify slow waves and time the sounds. Barely audible sounds are delivered through headphones and played during sleep (specifically, during slow wave sleep).
  Arms: MCI auditory stimulation; Older adult auditory stimulation
Other: Sham Intervention — The brain electroencephalogram is measured and headphones are worn, but sounds are not played during sleep.
  Arms: MCI sham stimulation; older adult sham stimulation

SUMMARY:
This study will evaluate the ability of sounds played during slow wave sleep using a phase locked loop algorithm to enhance slow wave sleep and memory in cognitively healthy older adults and in those with amnestic mild cognitive impairment.

DETAILED DESCRIPTION:
Alzheimer's disease is a degenerative disorder associated with aging and presents a significant human and financial burden. Amnestic mild cognitive impairment (aMCI) is a disorder of impaired memory and is a precursor to Alzheimer's disease. Current treatments are symptomatic and do not slow disease progression. There is increasing evidence linking sleep and cognition, such that decreased sleep, particularly slow wave sleep (physiologically slow wave activity; SWA), is associated with impaired cognitive performance. Not only does SWA decrease with aging, it is much less in people with aMCI than cognitively normal elderly. Interventions that improve sleep may also improve cognition. Auditory stimulation using sounds played through headphones or speakers during sleep have been shown to increase SWA and memory in young adults. Because this method plays sounds at fixed intervals, its ability to enhance SWA may be limited. Investigators have developed an improved method that measures slow waves during sleep in real time and delivers the sound at a particular phase of the slow wave (phase locked loop; PLL). Given that people with aMCI have low SWA, this method may be able to improve cognition by enhancing SWA. Our objective is to determine whether the PLL method of auditory stimulation can increase SWA and improve cognition in people with aMCI. Investigators propose a randomized sham-controlled cross-over study of auditory stimulation that population.

The specific aims are:

1. to determine a dose and duration of stimulation required to increase SWA by 10% in people with aMCI;
2. to determine the effect of the stimulus on cognitive performance in people with aMCI using word pair recall and the NIH Toolbox cognitive battery, which includes tests in multiple cognitive domains.

Investigators will recruit 15 participants with aMCI identified through the Northwestern University Cognitive Neurology and Alzheimer's Disease Center Clinical Core. Participants will undergo 2 separate nights of polysomnography (stimulation and sham) and cognitive testing on stimulation and sham visits. There will be approximately 1 week between overnight visits. The order of stimulation and sham will be randomized. Results study will be used to determine the optimal stimulation parameters, provide preliminary data on its potential effect, and guide design of future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age ≥60 years;
2. Amnestic MCI group: Diagnosis of aMCI based on change in cognition compared to the individual's previous level, impairment of episodic memory, preserved independence in functional abilities, and no evidence of impairment in social or occupational functioning;
3. Healthy Older Adults Group: Intact cognitive profile based on neuropsychology testing within 1 standard deviation for age and education status.
4. regular reported sleep and wake times

Exclusion Criteria:

1. moderate-severe sleep apnea defined by apnea-hypopnea index ≥15 events/hour or periodic limb movement index ≥15/hour on the screening home sleep test;
2. unstable medical or psychiatric disorder;
3. currently doing rotating shift work or night work;
4. history of seizures or taking medications that may lower the seizure threshold;
5. current use of any sedative/hypnotics or stimulants, gabapentin, pregabalin, tricyclic antidepressants, and trazodone or other psychoactive medications that may alter slow wave sleep; however, stable (3 months or longer) use of antidepressants will be allowed.
6. hearing loss

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Memory performance on a word pair recall | Through study completion, approximately 1.5 years.
  Participants will initially view word pairs on a computer screen. Participants then complete a recall, where they are presented with one word and freely recall the second word from the pair. Participants complete word pair recall prior to sleep and then again after waking in the morning. This test is completed during both experiment visits.

SECONDARY OUTCOMES:
NIH Cognition Toolbox - Composite score | Through study completion, approximately 1.5 years.
  Participants will complete the NIH toolbox in the morning following both experimental nights. The investigators are evaluating composite scores from the NIH Cognition Toolbox between the two nights.

CONTACTS AND LOCATIONS:
Overall Officials: Roneil G Malkani, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersen RC. Mild cognitive impairment as a diagnostic entity. J Intern Med. 2004 Sep;256(3):183-94. doi: 10.1111/j.1365-2796.2004.01388.x. PMID 15324362
- [Background] Born J, Rasch B, Gais S. Sleep to remember. Neuroscientist. 2006 Oct;12(5):410-24. doi: 10.1177/1073858406292647. PMID 16957003
- [Background] Mander BA, Rao V, Lu B, Saletin JM, Lindquist JR, Ancoli-Israel S, Jagust W, Walker MP. Prefrontal atrophy, disrupted NREM slow waves and impaired hippocampal-dependent memory in aging. Nat Neurosci. 2013 Mar;16(3):357-64. doi: 10.1038/nn.3324. Epub 2013 Jan 27. PMID 23354332
- [Background] Dijk DJ, Beersma DG, van den Hoofdakker RH. All night spectral analysis of EEG sleep in young adult and middle-aged male subjects. Neurobiol Aging. 1989 Nov-Dec;10(6):677-82. doi: 10.1016/0197-4580(89)90004-3. PMID 2628779
- [Background] Van Cauter E, Leproult R, Plat L. Age-related changes in slow wave sleep and REM sleep and relationship with growth hormone and cortisol levels in healthy men. JAMA. 2000 Aug 16;284(7):861-8. doi: 10.1001/jama.284.7.861. PMID 10938176
- [Background] Ngo HV, Claussen JC, Born J, Molle M. Induction of slow oscillations by rhythmic acoustic stimulation. J Sleep Res. 2013 Feb;22(1):22-31. doi: 10.1111/j.1365-2869.2012.01039.x. Epub 2012 Aug 23. PMID 22913273
- [Background] Tononi G, Riedner BA, Hulse BK, Ferrarelli F, Sarasso S. Enhancing sleep slow waves with natural stimuli. Medicamundi 2010;54:73-9.